CLINICAL TRIAL: NCT06559384
Title: Facilitators and Barriers to Dental Care in Head and Neck Cancer Patients - Perspectives From Patients, Dentists, and Oncologists
Brief Title: Facilitators and Barriers to Dental Care in Head and Neck Cancer Patients
Status: Completed | Type: Observational
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Felix Marschner, Principal Ivestigator, University Medical Center Goettingen
Other Study IDs: 2024-03239
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Behavior
Keywords: interviews; decision-making
MeSH Terms: conditions — Behavior | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- German Dentists: Dentists who are working in dental offices in Germany
  Interventions: Other: Interviews
- German Oncologists: Oncologists who are working in private practice/clinics in Germany
  Interventions: Other: Interviews
- Patients with head-neck cancer: Patients with head and neck cancer or after therapy for head and neck tumors
  Interventions: Other: Interviews

INTERVENTIONS:
Other: Interviews — semi-structured individual interviews

SUMMARY:
The aim of this study is to identify potential facilitators and barriers to dental care in head-neck cancer patients from the perspective of affected patients, dentists, and oncologists (specialists in radiotherapy and specialists in otolaryngology).

DETAILED DESCRIPTION:
Patients as well as dentists and oncologists will be interviewed in semi-structured individual interviews. The interview guide used will align with the 14 domains of the Theoretical Domains Framework. Through qualitative content analysis, both facilitators and barriers to dental treatment for head-neck cancer patients will be identified.

ELIGIBILITY:
Inclusion Criteria:

* Patients with head and neck tumors whose health condition allows for the conduction of an interview
* Dentists practicing in Germany
* Specialists in otorhinolaryngology practicing in Germany
* Specialists in radiation therapy practicing in Germany

Exclusion Criteria:

* Missing consent for the study
* Health condition that does not allow the conduction of an interview

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with head-neck cancer, dentists (general dentists and specialised dentists) who are working in clinics and private practices in Germany and oncologists (specialists in radiotherapy and specialists in otolaryngology) who are working in Germany
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Questionnaire | 5 minutes
  Completion of a questionnaire
Interview | 60 minutes
  Semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Felix Marschner, Dr., Principal Investigator — University Medical Center Goettingen, Department of Preventive Dentistry, Periodontology and Cariology
Locations (1):
- University Medical Center Göttingen, Göttingen, Germany